CLINICAL TRIAL: NCT06224153
Title: Assessment of Protein Intake Using 2 Types of Nutritional Collection in Comparison with 24-hour Urine Urea, in Chronic Kidney Disease.
Brief Title: Assessment of Protein Intake Using 2 Types of Nutritional Collection in Chronic Kidney Disease.
Acronym: APRONUT_MRC
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: RCAPHM22_0201; ID-RCB (Other: 2023-A00510-45)
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Chronic Kidney Disease (stages 4 and 5)
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Diet Records

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with chronic kidney disease
  Interventions: Other: 3-day dietary record; Other: Food Frequency Questionnaire (FFQ)

INTERVENTIONS:
Other: 3-day dietary record — This is the conventional ingesta assessment. It will be performed twice during the study.
Other: Food Frequency Questionnaire (FFQ) — This questionnaire is used to obtain information on the frequency of foods and drinks consumed over a period of time (1 week, 1 month...). It will be performed twice during the study.

SUMMARY:
In France, 10% of the population suffers from chronic kidney disease (CKD). CKD is classified into five stages, described from the least severe (stage 1) to the most severe (stage 5). Every year, in the PACA region, around 1,000 new patients present with end-stage CKD (5D), necessitating the introduction of suppletive therapy, whether hemodialysis, peritoneal dialysis or kidney transplantation. In CKD stages 4 and 5, a hypo-protein diet can be proposed to delay dialysis initiation (Garneata et al. 2016).

To introduce a low-protein diet, the dietician first assesses protein intake. This can be done by :

* Measuring 24-hour urine urea. This is the reference method for assessing the amount of protein consumed over the last 24 hours. However, it cannot be used to determine the patient's dietary habits, and therefore cannot be used to suggest modifications with a view to introducing a low-protein diet.
* A detailed dietary record. The 3-day dietary record currently in use (a tool for recording dietary habits defined by the HAS) provides a reliable assessment of protein intake. However, this tool takes up a lot of dietetic time, limiting the time available for nutrition education and the number of patients who can benefit from a dietetic consultation.

MS-Nutrition is a start-up that has developed a web application that can be used by patients themselves to assess nutritional intakes, incorporating a food frequency questionnaire (known as the FFQ questionnaire) used to obtain information on the frequency of foods and drinks consumed over a period of time (1 week, 1 month...).

For the general population (without CKD), there is good agreement between the FFQ questionnaire and a conventional ingesta assessment (3-day dietary record as currently practiced or 24h recall, another collection based on the previous day's consumption) (Affret et al., 2018; Deschamps et al., 2009). These studies on healthy adults do not take into account the reference method (urinary urea) for assessing protein intake.

Only one study in the CKD population evaluates the concordance of the assessment of protein intakes (as well as calcium, phosphorus, potassium and sodium intakes) between an FFQ questionnaire and a dietary record (24-hour recall) (Affret et al. 2017). This study shows an acceptable correlation between the FFQ and the dietary record (correlation coefficient between 0.05 and 0.79, with a median of 0.40), yet this study was carried out without dietary intervention and using a different type of dietary record. As in studies on a population of healthy adults, protein intakes assessed by any type of dietary questionnaire are not compared with a more reliable assessment of these same intakes (24-hour urine urea).

The proposed study will compare the concordance of dietary intake assessment between each of the 2 types of dietary collection (FFQ and a 3-day dietary collection) and 24-hour urine urea, which limits the biases inherent in dietary collection.

ELIGIBILITY:
Inclusion Criteria:

* Patient at least 18 years of age,
* Patient capable of understanding the study and having given informed non-opposition,
* Patient with stage 4 or 5 CKD,
* Patient included in the MRC pathway,
* Patient motivated by a hypo-protein diet,
* Patient able to use a computer/smartphone/tablet with Internet access.

Exclusion Criteria:

* Difficulty reading or understanding the French language,
* Patient with ongoing cancer,
* Patient undernourished or at risk of undernutrition (based on weight loss and albumin measurement from last blood test),
* Persons covered by articles L. 1121-5 to L. 1121-8 of the French Public Health Code (minors, adults under guardianship or trusteeship, patients deprived of their liberty, pregnant or breast-feeding women).
* Dialysis patient
* Patient who underwent major surgery less than 3 months ago.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidney disease at stage 4 ou 5
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Estimation of the concordance between the reference method (24-hour urinary urea) and : (1) protein intake estimated by the 3-day dietary record ; (2) protein intakes estimated by FFQ via web application at the initial dietary consultation. | Between 15 days and 1 month

SECONDARY OUTCOMES:
Assessment of concordance between protein intake estimated by the 3-day dietary record and 24-hour urine urea measurement 6 months after the initial dietary consultation | Between 6 and 7 months
Assessment of concordance between protein intakes estimated by FFQ via web application and 24-hour urine urea measurement 6 months after the initial dietary consultation | Between 6 and 7 months
Evaluation and comparison of the time taken by the dietician to collect the data required to assess protein intake with the 2 types of dietary record at the initial dietary consultation | Between 15 days and 1 month
Evaluation and comparison of the time taken by the dietician to collect the data required to assess protein intake with the 2 types of dietary record 6 months after the initial dietary consultation | Between 6 and 7 months
Assessment of the concordance between nutritional intakes obtained by the 2 food collection methods at the initial dietary consultation | Between 15 days and 1 month
Assessment of the concordance between nutritional intakes obtained by the 2 food collection methods 6 months after the initial dietary consultation | Between 6 and 7 months

CONTACTS AND LOCATIONS:
Overall Officials: François CREMIEUX, Study Director — AP-HM
Locations (1):
- Centre de néphrologie et de transplantation rénale, Marseille, France, France

IPD SHARING:
Plan to Share IPD: Undecided